CLINICAL TRIAL: NCT02312401
Title: Evaluation of Treatment Response Using Multiparametric MRI After Prostate Radiotherapy
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-172
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: MRI; 14-172
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dynamic Contrast Enhanced Magnetic Resonance Imaging; Biopsy

ARMS (1):
- Multiparametric MRI (Experimental): Patients undergo baseline standard (clinical) MP-MRI prior to therapy (ADT or RT). After completion of radiotherapy, follow-up MRIs will be obtained using the same 3T Philips MRI unit at approximately 3, 6, 12, 18 & 24 (+/- 4 weeks) months after radiotherapy. A standard post-tx biopsy will be performed at 24 months (+/- 4 weeks) after therapy which will serve to define the local control status after therapy. Local control based on this biopsy will be interpreted as negative or adenoca with severe tx effect; a positive biopsy will be a specimen which demonstrates adenocarcinoma that can be classified with a Gleason score as we have previously reported.
  Interventions: Device: multi-parametric MRI(MP-MRI); Device: dynamic contrast-enhanced MRI (DCE); Procedure: biopsy

INTERVENTIONS:
Device: multi-parametric MRI(MP-MRI)
Device: dynamic contrast-enhanced MRI (DCE)
Procedure: biopsy

SUMMARY:
The purpose of this study is to better understand prostate cancer changes after radiation treatment, through magnetic resonance imaging (MRI). MRI is an imaging test that allows doctors to see prostate gland without any operation procedures. It can help identifying the tumors in the prostate. For patients with newly diagnosed prostate cancer, MRI may help doctors manage treatment better and sooner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with biopsy proven (completed and/or reviewed at MSK) adenocarcinoma of the prostate, who will undergo external beam radiotherapy using conventional fractionation IGRT including moderate hypofractionated radiation, low rate brachytherapy alone, brachytherapy (either high dose or low dose) combined with supplemental image guided radiation (including IGRT, EBRT, and SBRT), SBRT, or proton radiotherapy.
* Age ≥ 18 years old
* Baseline MP-MRI, which is obtained at MSKCC Main Campus on the 3-Tesla Philips MRI unit as part of the standard (clinical) staging assessment demonstrates at least one dominant or visible lesion which measures > 0.5 cm in maximum axial diameter as assessed on T2-weighted images.
* No prior history of androgen deprivation therapy within the last month. However patients who will receive neoadjuvant and concurrent and adjuvant hormonal therapy will be eligible.
* Willing to come to MSK Main Campus for baseline and follow-up MP-MRIs.

Exclusion Criteria:

* History of radical prostatectomy
* Patients who are unwilling or unable to undergo MRI including patients with contraindications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips, claustrophobia, inability to lie flat for the duration of the study etc.
* Patients with a metallic hip implant, metallic implant or device in the pelvis or ferromagnetic fiducial beacons (Calypso) that might distort local magnetic field and compromise quality of MP-MRI
* Patients in which gadolinium contrast is contra-indicated.
* Metastatic disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
characterize the changes in tumor characteristics by functional imaging changes with post-treatment prostate biopsy outcomes | at 24 months after completion of radiotherapy
  This change will then be correlated with the biopsy outcome (binary) by two sample t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Neelam Tyagi, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Rockville Centre, Rockville Centre, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/